CLINICAL TRIAL: NCT03873051
Title: Developing Real Incentives and Volition for Exercise Project
Brief Title: Developing Real Incentives and Volition for Exercise
Acronym: DRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Allison M. Sweeney, Postdoctoral Fellow, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00085166; F32HL138928-01A1 (NIH)
Record Dates: First submitted 2019-03-02; First posted 2019-03-13 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity
Keywords: Community-based intervention; Motivation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The randomized pilot study compares the effects of receiving a matched (Autonomous & Challenge-Focused; Controlled & Rewards-Focused) versus an non-matched (Autonomous & Rewards-Focused; Controlled & Challenge -Focused) group-based PA intervention program over an 8-week time period. Randomization to the Rewards- or Challenge-focused intervention is stratified by degree of autonomous motivation (low, medium, high). A total of 150 African American women will be randomly assigned to either receive the Rewards- or the Challenge-focused intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Challenge-Focused Program (Experimental): This group will receive the challenge-focused group program
  Interventions: Behavioral: Challenge-Focused Program
- Rewards-Focused Program (Experimental): This group will receive the rewards-focused group program
  Interventions: Behavioral: Rewards-Focused Program

INTERVENTIONS:
Behavioral: Challenge-Focused Program — Participants receiving the Challenge-Focused intervention will complete an 8-week group program. Group sessions meet once per week for 90 minutes and include three components - discussion-based health promotion initiative, team-based physical activity games/activities, and team-based goal-setting and behavioral skills training. Among participants with high autonomous motivation, those receiving the Challenge-focused intervention are expected to show greater improvement from baseline to post- in total PA than those receiving the Rewards-Focused intervention.
  Arms: Challenge-Focused Program
Behavioral: Rewards-Focused Program — Participants receiving the Rewards-Focused intervention will complete an 8-week group program. Group sessions meet once per week for 90 minutes and include three components - discussion-based health promotion initiative, group-based walking program, and individual-based goal-setting and behavioral skills training with partner-based contracts and financial incentives. Among participants with high controlled motivation, those receiving the Rewards-focused intervention are expected to show greater improvement from baseline to post- in total PA than those receiving the Challenge-Focused intervention.
  Arms: Rewards-Focused Program

SUMMARY:
The overall goal of the Developing Real Incentives and Volition for Exercise (DRIVE) Project is to evaluate whether matching an intervention to individual differences in motivation (high autonomous vs high controlled) is a feasible strategy for engaging African American women in greater total physical activity (PA). The DRIVE Project will develop and evaluate two novel interventions: 1) a challenge-focused program that targets greater PA enjoyment, PA valuation, and relatedness through team-based activities, behavioral skills, and a positive social climate; and 2) a rewards-focused program that targets greater PA competency and relatedness through financial incentives, behavioral skills, and structured social support. To this end, the investigators will be implementing a randomized pilot study at a community center. It is hypothesized that participants who receive an intervention that is matched to their motivation for PA initiation (High Autonomous & Challenge-Focused; High Controlled & Rewards-Focused) will demonstrate greater improvements from baseline to post- in total physical activity than those who receive an unmatched intervention (High Autonomous & Rewards-Focused; High Controlled & Challenge-Focused). The DRIVE project will provide proof-of-concept for the feasibility and usefulness of developing motivationally-targeted intervention programs for engaging African American women in greater PA.

DETAILED DESCRIPTION:
Although engaging in regular physical activity (PA) plays a critical role in reducing one's risk for numerous health problems, 4 out of 5 U.S. adults fail to meet national PA guidelines, with underserved groups (low income and racial/ethnic minority groups) having the highest rates of physical inactivity. Developing innovative strategies to motivate underserved groups to initiate PA has become an increasing national priority, but many implementation challenges remain, as evidenced by relatively low levels of program engagement among underserved groups. Increasingly, researchers have begun to show that rather than using a "one-size-fits all" intervention approach, developing interventions that target specific individual differences in cultural or social-cognitive factors is a highly effective approach for increasing engagement among underserved groups. Broadening this approach in a novel domain, the proposed research tests whether developing interventions that target differences in autonomous (internally-driven) vs. controlled (externally-driven) motivation is a feasible and useful approach for engaging African American women in PA initiation. The proposed study is a randomized pilot study comparing two intervention programs: a Challenge-focused program targeted toward high autonomous motivation and a Rewards-focused program targeted toward high controlled motivation. The Challenge-focused program targets greater PA enjoyment, PA valuation, and relatedness, and the Rewards-focused program targets greater PA competence and structured social support for PA. It is hypothesized that baseline motivation (measured with the Behavioral Regulation in Exercise questionnaire) will moderate treatment effects. Specifically, participants with relatively higher autonomous motivation will demonstrate greater improvements from baseline to post- in total physical activity when they receive the "matched" intervention (Challenge-Focused program) relative to the non-matched intervention (Rewards-Focused Program). Additionally, participants with relatively higher controlled motivation will demonstrate greater improvements from baseline to post- in total physical activity when they receive the "matched" intervention (Rewards-Focused program) relative to the non-matched intervention (Challenge-Focused Program). The results of this study will provide support of the feasibility and proof-of-concept for conducting a large scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Female
* At least 21 years old
* Engage in < 150 min. of moderate to vigorous physical activity per week for the last 3 months

Exclusion Criteria:

* Having a condition that would limit participation in PA (assessed with the Physical Activity Readiness Questionnaire)
* Uncontrolled blood pressure (> 180/120 mm Hg).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in total physical activity | Baseline to 2 months
  Average minutes of total physical activity (PA) per day; Objective assessments of total PA will be obtained with omni- directional accelerometers. Participants will wear the monitor affixed by an elastic belt over the right hip for 7 consecutive days during baseline and post-intervention (2 months). Consistent with previous studies, a valid day will consist of 10 hours of wear time, and 60 consecutive zeros will indicate non-wear with the allowance of up to 2 minutes under the count threshold for sedentary activity. Data reduction will use previously established accelerometer cut-points (Light PA: 100-1534, MVPA > = 1535), which will be summed to calculate total PA.

SECONDARY OUTCOMES:
Change in moderate to vigorous physical activity | Baseline to 2 months
  Average minutes of moderate to vigorous physical activity (MVPA) per day; Objective assessments of MVPA will be obtained with omni-directional accelerometers. Participants will wear the monitor affixed by an elastic belt over the right hip for 7 consecutive days during baseline and post-intervention (2 months). Consistent with previous studies, a valid day will consist of 10 hours of wear time, and 60 consecutive zeros will indicate non-wear with the allowance of up to 2 minutes under the count threshold for sedentary activity. Data reduction will use previously established accelerometer cut-points, such that MVPA > = 1535.

OTHER OUTCOMES:
Change in Self-Efficacy for physical activity | Baseline to 2 months
  The Self-Efficacy for Exercise Questionnaire (10 items; 5 point scale; 1-not at all confident; 5=extremely confident) will be used to evaluate self-efficacy for PA at baseline and 2 months (adapted from Sallis et al, 1988).
Change in Self-Concept for PA | Baseline to 2 months
  The Self Concept and Motivation to Exercise Scale (10 items; 1-strongly disagree, 6-strongly agree) will be used to evaluate self-concept for PA at baseline and 2 months (Wilson et al., 2002)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make the data (psychosocial, physical activity, data dictionaries) available through a private study registration on the Open Science Framework. Study protocols, measures, and materials will also be made available on the the Open Science Framework. The PI will review requests for accessing the private study registration.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available after the primary and secondary outcome papers have been published (starting 6 months after publication).
Access Criteria: Requests will be reviewed by the PI, Allison Sweeney (sweeneam@mailbox.sc.edu). Requests must include information about the reason for wanting to access the data/materials and planned analyses.